CLINICAL TRIAL: NCT05671627
Title: An Impaired Functional Reserve of Adrenal Cortex May Associate With difficult-to Treat RA: Can a Disturbed Cortisol Circadian Rhythm Serve as a Predictor of Difficult-to-treat RA?
Brief Title: Cortisol Circadian Rhythm in Patients With RA
Acronym: CortRyRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maria Yavropoulou, Principal investigator, National and Kapodistrian University of Athens
Other Study IDs: EΣ-38/ 21-1-2021
Record Dates: First submitted 2022-09-19; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis
Keywords: salivary cortisol; hypothalamus-pituitary-adrenal axis; circadian rhythm; adrenals; response to treatment
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with Rheumatoid arthritis and good response at 3/6/12 months: Patients with Rheumatoid arthritis that fulfill the inclusion/exclusion criteria and show a good response at 3/6 or 12 months upon recruitment according to EULAR guidelines with or without corticosteroids (corticosteroid regimens do not exceed 15 mg/day) Patients will be treated as per clinician's judgement with any kind or combination of DMARDs with or without corticosteroids (corticosteroid regimens do not exceed 15 mg/day), following EULAR recommendations for RA treatment.
  Interventions: Drug: DMARDs
- patients with Rheumatoid arthritis and none at 3/6/12 months: Patients with Rheumatoid arthritis that fulfill the inclusion/exclusion criteria and show none response at 3/6 or 12 months upon recruitment according to EULAR guidelines.
  Patients will be treated as per clinician's judgement with any kind or combination of DMARDs with or without corticosteroids (corticosteroid regimens do not exceed 15 mg/day), following EULAR recommendations for RA treatment.
  Interventions: Drug: DMARDs

INTERVENTIONS:
Drug: DMARDs — Patients will be treated as per clinician's judgement with any kind or combination of DMARDs with or without corticosteroids (corticosteroid regimens do not exceed 15 mg/day), following EULAR recommendations for RA treatment.
  Other Names: Corticosteroid regimens that do not exceed 15 mg/day

SUMMARY:
The European League Against Rheumatism (EULAR), acknowledging the critical issue of the complications, of long term treatment with glucocorticoids in the most recent update of the management guidelines for Rheumatoid arthritis, recommends tapering (on sustained clinical remission) of oral glucocorticoids treatment at the earliest feasible time point of therapeutic course and to the lowest daily dose, preferably <7.5mg/day (prednisone equivalent), until the final target of withdrawal is succeeded. In clinical practice, these guidelines are often difficult to follow due to the high risk of disease flares after tapering or stopping glucocorticoids administration. This inability of tapering oral glucocorticoids below 7.5mg/day of prednisone or an equivalent synthetic glucocorticoid is included in the recent definition of difficult-to-treat Rheumatoid arthritis. SΕΜΙRΑ (Steroid EliMination In Rheumatoid Arthritis) study, a double-blind, multicentre, randomised controlled trial, compared oral glucocorticoids tapering with the continuation of low dose oral glucocorticoids. The population study consisted of 259 RA patients with low disease activity on treatment with 5mg per day prednisone and tocilizumab, an anti-interleukin (IL)-6 receptor antibody. The study demonstrated that the continued-prednisone regimen provided better maintenance of disease remission than did the tapered-prednisone regimen for the study period of 24 weeks with no symptoms suggestive of AI. However, the study protocol did not include biochemical assessment of adrenocortical function.

Experimental and clinical data have suggested that inadequate production of endogenous cortisol relative to enhanced clinical needs associated with the systemic inflammatory response, coined as the 'disproportion principle', may operate in Rheumatoid arthritis. Although the underlying molecular mechanisms remain unknown, both chronic overexpression of proinflammatory cytokines and chronic stress may contribute in the hyporesponsiveness of the hypothalamic-pituitary-adrenal axis and the target tissue glucocorticoid resistance that have been described, but not systematically studied. Thus, a precise longitudinal assessment of endogenous cortisol production may be needed for optimal management of patients with Rheumatoid arthritis. Based on the above, the investigators seek to investigate the hypothesis that an impaired functional reserve of adrenal cortex, due to chronic over-expression of pro-inflammatory cytokines and/or chronic stress may contribute to the development of Rheumatoid arthritis and/or associate with difficult-to treat RA. If this is the case, then a disturbed cortisol circadian rhythm reflecting this impairment may serve as a predictor of difficult-to-treat RA during the first diagnosis. In order to address this issue, the investigators designed a prospective cohort study including adult patients with Rheumatoid arthritis who require drug treatment for the first time or escalation of existing treatment due to active disease. Patients will be treated as per clinician's judgement with any kind or combination of DMARDs with or without corticosteroids (corticosteroid regimens when started will not exceed 15 mg/day, and will be given for at least 3 months), following EULAR recommendations for RA treatment.

Patients will be monitored at baseline, 3 months, 6 months and 12 months, assessing disease response to treatment, the need for continuing glucocorticoid treatment, inflammatory indexes, and diurnal salivary cortisol levels. Patients' classification will be based on EULAR response to treatment criteria for RA and cortisol circadian rhythm will be comparatively assessed (at baseline and at 3/6/12 months) between groups based on treatment response (EULAR guidelines).

DETAILED DESCRIPTION:
It is well known that a proportion of patients with RA is always in need of even small doses of glucocorticoids to maintain clinical remission, despite concomitant treatment with conventional and biologic disease-modifying drugs (DMARDs).The European League Against Rheumatism (EULAR), acknowledging the critical issue of the GCs-induced complications, suggested in the most recent update of the RA management guidelines tapering (on sustained clinical remission) of oral GCs treatment at the earliest feasible time point of therapeutic course and to the lowest daily dose, preferably <7.5mg/day (prednisone equivalent), until the final target of withdrawal is succeeded. In clinical practice, these guidelines are often difficult to follow. In any case, the inability of tapering oral GC below 7.5mg/day of prednisone or an equivalent synthetic GC is included in the recent definition of difficult-to-treat RA.

Experimental and clinical data have suggested that inadequate production of endogenous cortisol relative to enhanced clinical needs associated with the systemic inflammatory response, coined as the 'disproportion principle', may operate in RA. Although the underlying molecular mechanisms are unknown, both chronic overexpression of proinflammatory cytokines and chronic stress may contribute the most in the hyporesponsiveness of the hypothalamic-pituitary-adrenal axis and the target tissue glucocorticoid resistance that have been described, but not systematically studied. Thus, a precise longitudinal assessment of endogenous cortisol production may be needed for optimal RA management.

Recently the investigators have assessed the cortisol circadian rhythm, using saliva measurements, in patients with acute viral infection, as is COVID-19, comparing to healthy controls. In this study COVID-19 patients had almost 6-fold higher mean serum CRP and IL-6 levels than controls (p<0.001), whereas morning salivary cortisol levels were similar in the two groups. Diurnal cortisol rhythm in these patients was blunted, with increased evening and nocturnal levels, resulting in higher time-integrated daily cortisol secretion in patients than controls (area under the curve: 4.81±2.46 vs.2.75±0.810, respectively, p<0.001).

Based on the above, the investigators will test the hypothesis that an impaired functional reserve of adrenal cortex, due to chronic over-expression of pro-inflammatory cytokines and/or chronic stress may contribute to RA development and/or associate with difficult-to treat RA. If this is the case, then a disturbed cortisol circadian rhythm reflecting this impairment may serve as a predictor of difficult-to-treat RA.

In order to address this issue, the investigators designed the following study, considering the fact that the tested hypothesis seems to be a JANUS hypothesis since those patients who are at need of corticosteroids to maintain low disease activity or remission could have either high or low evening/night cortisol levels at baseline.

Study Design

This is a single-center prospective cohort study of 50 consecutive RA adult patients (fulfilling the 2010 ACR/EULAR classification criteria) who are:

1. newly -diagnosed and are going to start treatment, or
2. require escalation of drug treatment due to active disease (addition of biologic or cDMARD or change of biologic with or without corticosteroids) providing that are off corticosteroid treatment for at least 3 months.

Patients will be treated as per clinician's judgement with any kind or combination of DMARDs with or without corticosteroids (corticosteroid regimens do not exceed 15 mg/day), following EULAR recommendations for RA treatment.

Time points of assessment:

Baseline (day 0), months 3, months 6 and 12 months. Blood samples, diurnal salivary cortisol samples and questionnaires regarding self-perceived stress and Hamilton scale for depression will be collected from all recruited individuals. Important NOTE: those who are on corticosteroids at 3 and/or 6 months (preferably below 7.5mg of prezolon) will be advised to stop corticosteroids treatment for 48 h before saliva measurements.

Patients' classification will be based on EULAR response to treatment criteria for RA at month 3 and month 6 and 12 months compared to baseline (moderate and good response patients may be considered together).

Patients will be recruited from the Outpatient clinic for Rheumatology and autoimmune diseases of Medical School, National and Kapodistrian University of Athens located at LAIKO University Hospital, 17 Agiou Thoma, 11527, Athens, Greece.

Cortisol circadian rhythm will be comparatively assessed (at baseline and at 3/6/12 months) between responders Vs non-responders and a post-hoc analysis will be performed on the longitudinal changes in the cortisol circadian rhythm in relation to the clinical status and stress/depression levels of the individual patients.

Age- and sex-matched apparently healthy volunteers who fulfill the inclusion/exclusion criteria will be recruited from the Hospital personnel during the same time-period and serve as controls, in a case -control, cross-sectional analysis to investigate differences between circadian cortisol rhythm between patients and healthy individuals.

All participants will sign an informed consent and the procedures followed will be in accordance with the 1975/83 Declaration of Helsinki. The study is approved by the scientific committee of Laikon Athens University-Hospital (Approval number E.Σ. 38/21-01-2021).

ELIGIBILITY:
Inclusion Criteria:

RA adult patients (fulfilling the 2010 ACR/EULAR classification criteria) who are:

1. Newly -diagnosed and are going to start treatment, or
2. require escalation of drug treatment due to active disease (addition of biologic or cDMARD or change of biologic with or without corticosteroids) providing that are off corticosteroid treatment for at least 6 months.

Exclusion Criteria:

* chronic kidney disease stage 3b and above,
* antineoplastic treatment,
* TSH>10 IU/lt,
* Cushing syndrome
* hypo-/hyper-parathyroidism
* estrogen replacement therapy
* insulin treatment or HBA1c>7.5 %,
* BMI>35
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients fulfilling the 2010 ACR/EULAR classification criteria that visit the Outpatient clinic for Rheumatology and autoimmune diseases.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Circadian Rhythm of cortisol | Salivary samples will be obtained at prescheduled timepoints, 8am, for measurement of free cortisol levels.
  Salivary samples for cortisol measurements will be collected using the Salivette device (Sarstedt, Nümbrecht, Germany). The participants will be asked to refrain from eating and brushing their teeth for 1 hour before the collection. The measurements will be performed by an electrochemiluminescence immunoassay on the automated analyzer Cobas e411-Roche Diagnostics (GmbH, Mannheim). The detection limit is 0.054 mcg/dL and the intra- and inter-assay CV is 6.1% and 11.8%, respectively, at the concentration of 0.137 mcg/dL.
Circadian Rhythm of cortisol | Salivary samples will be obtained at 12-noon for measurements of free cortisol levels.
  Salivary samples for cortisol measurements will be collected using the Salivette device (Sarstedt, Nümbrecht, Germany). The participants will be asked to refrain from eating and brushing their teeth for 1 hour before the collection. The measurements will be performed by an electrochemiluminescence immunoassay on the automated analyzer Cobas e411-Roche Diagnostics (GmbH, Mannheim). The detection limit is 0.054 mcg/dL and the intra- and inter-assay CV is 6.1% and 11.8%, respectively, at the concentration of 0.137 mcg/dL.
Circadian Rhythm of cortisol | Salivary samples will be obtained at 6pm for measurements of free cortisol levels.
  Salivary samples for cortisol measurements will be collected using the Salivette device (Sarstedt, Nümbrecht, Germany). The participants will be asked to refrain from eating and brushing their teeth for 1 hour before the collection. The measurements will be performed by an electrochemiluminescence immunoassay on the automated analyzer Cobas e411-Roche Diagnostics (GmbH, Mannheim). The detection limit is 0.054 mcg/dL and the intra- and inter-assay CV is 6.1% and 11.8%, respectively, at the concentration of 0.137 mcg/dL.
Circadian Rhythm of cortisol | Salivary samples will be obtained at 10pm for measurements of free cortisol levels.
  Salivary samples for cortisol measurements will be collected using the Salivette device (Sarstedt, Nümbrecht, Germany). The participants will be asked to refrain from eating and brushing their teeth for 1 hour before the collection. The measurements will be performed by an electrochemiluminescence immunoassay on the automated analyzer Cobas e411-Roche Diagnostics (GmbH, Mannheim). The detection limit is 0.054 mcg/dL and the intra- and inter-assay CV is 6.1% and 11.8%, respectively, at the concentration of 0.137 mcg/dL.

SECONDARY OUTCOMES:
Serum DHEAS levels | Blood samples will be obtained from patients and controls immediately upon recruitment at morning hours after overnight fast
  Measurement of DHEAS levels (Immulite 2000 Siemen)
Serum DHEAS levels | Blood samples will be obtained from patients at 3 months of treatment during morning hours after overnight fast
  Measurement of DHEAS levels (Immulite 2000 Siemen)
Serum DHEAS levels | Blood samples will be obtained from patients at 6 months of treatment during morning hours after overnight fast
  Measurement of DHEAS levels (Immulite 2000 Siemen)
Serum DHEAS levels | Blood samples will be obtained from patients at 12 months of treatment during morning hours after overnight fast
  Measurement of DHEAS levels (Immulite 2000 Siemen)
Plasma ACTH levels | Blood samples will be obtained from patients and controls immediately upon recruitment at morning hours after overnight fast
  Measurement of morning plasma ACTH levels sing solid-phase, two-site chemiluminescence immunoassays on an IMMULITE 2000 Immunoassay System (Siemens Healthcare Diagnostics Products Ltd, UK). ). The analytical sensitivity for ACTH measurement is 5 pg/mL . . The intra and inter- assay coefficients of variation (CV) for ACTH ranges from 6.7 to 9.5 % and from 6.1 to 10 %, respectively
Serum CRP levels | Blood samples will be obtained from patients and controls immediately upon recruitment at morning hours after overnight fast
  Serum high sensitivity CRP (hsCRP) will be measured using solid-phase, two-site chemiluminescence immunoassays on an IMMULITE 2000 Immunoassay System (Siemens Healthcare Diagnostics Products Ltd, UK). The analytical sensitivity for hsCRP measurement is 0.1 mg/L. The intra and inter- assay coefficients of variation (CV) for hsCRP from 2.8 to 8.7 % and from 3.1 to 8.7 %, respectively, depending on the sample concentration.
Serum IL-6 levels | Blood samples will be obtained from patients and controls immediately upon recruitment at morning hours after overnight fast
  Measurement of IL-6 levels was detected by a sandwich enzyme immunoassay using Quantikine ELISA kit (R&D Systems, Minneapolis, MN, USA). The lower detection limit of DIAsource aldosterone assay is 15 pg/mL and the intra- and inter- assay CV lays between 4.5 and 8.7 %, respectively, depending on sample concentration. The lower detectable measurement of IL-6 is 0.70 pg/mL and the inter- and intra- assay precision ranged between 1.6 and 4.2 and from 3.3 to 6.4, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Laiko General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yavropoulou MP, Filippa MG, Panopoulos S, Spanos E, Spanos G, Tektonidou MG, Sfikakis PP. Impaired adrenal cortex reserve in patients with rheumatic and musculoskeletal diseases who relapse upon tapering of low glucocorticoid dose. Clin Exp Rheumatol. 2022 Sep;40(9):1789-1792. doi: 10.55563/clinexprheumatol/x78tko. Epub 2022 Jun 13. PMID 35699085
- [Background] Tan Y, Buch MH. 'Difficult to treat' rheumatoid arthritis: current position and considerations for next steps. RMD Open. 2022 Jul;8(2):e002387. doi: 10.1136/rmdopen-2022-002387. PMID 35896282
- [Background] Burmester GR, Buttgereit F, Bernasconi C, Alvaro-Gracia JM, Castro N, Dougados M, Gabay C, van Laar JM, Nebesky JM, Pethoe-Schramm A, Salvarani C, Donath MY, John MR; SEMIRA collaborators. Continuing versus tapering glucocorticoids after achievement of low disease activity or remission in rheumatoid arthritis (SEMIRA): a double-blind, multicentre, randomised controlled trial. Lancet. 2020 Jul 25;396(10246):267-276. doi: 10.1016/S0140-6736(20)30636-X. PMID 32711802
- [Background] Yavropoulou MP, Filippa MG, Mantzou A, Ntziora F, Mylona M, Tektonidou MG, Vlachogiannis NI, Paraskevis D, Kaltsas GA, Chrousos GP, Sfikakis PP. Alterations in cortisol and interleukin-6 secretion in patients with COVID-19 suggestive of neuroendocrine-immune adaptations. Endocrine. 2022 Feb;75(2):317-327. doi: 10.1007/s12020-021-02968-8. Epub 2022 Jan 18. PMID 35043384
- [Background] Smolen JS, Landewe R, Breedveld FC, Dougados M, Emery P, Gaujoux-Viala C, Gorter S, Knevel R, Nam J, Schoels M, Aletaha D, Buch M, Gossec L, Huizinga T, Bijlsma JW, Burmester G, Combe B, Cutolo M, Gabay C, Gomez-Reino J, Kouloumas M, Kvien TK, Martin-Mola E, McInnes I, Pavelka K, van Riel P, Scholte M, Scott DL, Sokka T, Valesini G, van Vollenhoven R, Winthrop KL, Wong J, Zink A, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2010 Jun;69(6):964-75. doi: 10.1136/ard.2009.126532. Epub 2010 May 5. PMID 20444750
- [Background] Fransen J, van Riel PL. The Disease Activity Score and the EULAR response criteria. Rheum Dis Clin North Am. 2009 Nov;35(4):745-57, vii-viii. doi: 10.1016/j.rdc.2009.10.001. PMID 19962619
- [Derived] Yavropoulou MP, Filippa MG, Vlachogiannis NI, Fragoulis GE, Laskari K, Mantzou A, Panopoulos S, Fanouriakis A, Bournia VK, Evangelatos G, Papapanagiotou A, Tektonidou MG, Chrousos GP, Sfikakis PP. Diurnal production of cortisol and prediction of treatment response in rheumatoid arthritis: a 6-month, real-life prospective cohort study. RMD Open. 2024 Jan 17;10(1):e003575. doi: 10.1136/rmdopen-2023-003575. PMID 38233075